CLINICAL TRIAL: NCT07275866
Title: A Pilot Study of a Multi-Strain Liquid Probiotic in Individuals Self-reporting Constipation in the General Population.
Brief Title: Multi-strain Probiotic Effects on Self-Reported Constipation
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Dr Anthony Hobson (Other)
Responsible Party: Sponsor-Investigator, Dr Anthony Hobson, Clinical Director and Senior Clinical GI Scientist, The Functional Gut Clinic
Organization: The Functional Gut Clinic (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FGC-25-02
Record Dates: First submitted 2025-11-27; First posted 2025-12-10 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-11

CONDITIONS: Constipation; Probiotic; Probiotic Intervention
MeSH Terms: conditions — Constipation

STUDY DESIGN:
Intervention Model Description: The study is a single arm open label treatment. The study comprises of a 2 week baseline period followed by a 4 week treatment period.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Multi-strain Liquid Probiotic (Experimental): 70ml of a multi-strain liquid probiotic taken daily for 28-35 days
  Interventions: Dietary Supplement: Multi-strain probiotics

INTERVENTIONS:
Dietary Supplement: Multi-strain probiotics — 28-35 days of 70 ml Symprove once daily, to be taken on an empty stomach upon waking. 10 minutes should be taken between ingestion of Symprove before eating and drinking.

SUMMARY:
Constipation is a prevalent gastrointestinal condition. Beyond simple lifestyle measures (e.g. increasing fibre intake, hydration, levels of exercise), medical therapies are available for management. However, a sizeable number of sufferers are dissatisfied with drug treatments (either over-the-counter or prescribed), meaning there is an unmet need for alternative therapeutic strategies.

Pre, pro- and synbiotics have emerged as one alternative treatment, and a growing body of evidence now supports their use in a proportion of individuals with mild constipation. However, it is currently not possible to predict which individuals may benefit. A better understanding of an individuals' symptoms and underlying pathophysiology may allow for more targeted treatment.

The multistrain live bacterial food product (probiotic) being tested contains billions of live and active bacteria that has been shown to improve symptoms in the irritable bowel syndrome (IBS: which is 'constipation-predominant' in many). Notably, improvements ('completely resolved' or 'some positive difference') in bowel habit satisfaction, abdominal pain, bloating and urgency, as well as on quality of life have been shown after 4 or more weeks of this probiotc.

This study aims to have 20 participants with self-reported constipation to assess improvements in constipation symptoms, quality of life and measures of gut function.

ELIGIBILITY:
Inclusion Criteria:

1. Participant has provided written informed consent before participating in the study after being given a full description of the study and prior to any study-specific procedures being performed.
2. Participant has Cleveland Clinic constipation score (CCCS) of 9-16 at screening call
3. Participant is willing to discontinue all other therapies for constipation and undergo washout where applicable.
4. Participant is a male or non-pregnant female and is 18-70 years of age
5. If WOCBP participant is willing to adhere to one of the following methods of contraception:

   i) Hormonal contraception e.g. the 'pill' or an implant ii) Intrauterine device (IUD) iii) Intrauterine hormone-releasing system (IUS) vi) Sexual abstinence (if it is in line with participants' preferred and usual lifestyle).

   or has had a: v) Hysterectomy or has a: vi) Vasectomised partner
6. Participant can communicate well with the Investigator and to comply with the requirements for the entire study.
7. Participant has capacity to understand written English.
8. Participant has a body mass index (BMI) of 18.5 - 39.9kg/m2 (bounds included).
9. Participant agrees to follow all pre-test preparation for the ATMO capsule transit study.

Exclusion Criteria:

1. Women who are pregnant and/or breastfeeding.
2. Participants who are planning to significantly change their diet (e.g. weight loss program, becoming vegetarian) during the study period.
3. Participant has had diarrhoea within 7 weeks of screening period.
4. Prior abdominal surgery involving resection of the small or large bowel.
5. Prior bariatric surgery involving resection of the stomach or by-pass procedures.
6. Type 1 diabetes mellitus.
7. Known organic or structural GI disease including:

   * Coeliac disease
   * Inflammatory bowel disease
   * Diverticulitis
   * Small bowel strictures
8. Irritable bowel syndrome where the predominant symptom is pain (assessed via screening questions).
9. Oropharyngeal dysphagia or difficulty swallowing capsules.
10. Any other medical condition that the investigator deems may confound results or affect participants' safety in the study.
11. Any use of prohibited medication that the participant cannot complete appropriate washout for.
12. Insufficient knowledge of English to complete the daily bowel diary.
13. Allergy to any component of the supplement, motility bar, lactulose or Zoe blue cookie.
14. Participant is involved in this study as an investigator, sub-Investigator, study coordinator, other study staff, or Sponsor member.
15. Previous use of the probiotic Symprove.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-10-03 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Patient Assessment of Constipation-Symptoms (PAC-SYM) | Pre-post comparison (28 days)
  Number of participants with clinically meaningful change in PAC-SYM score (reduction of >0.6 or >0.75 points).
  The PAC-SYM questionnaire is a 12 item validated patient-reported measure of severity of constipation symptoms during the past two weeks.

SECONDARY OUTCOMES:
Patient Assessment of Constipation - Quality of Life (PAC-QoL) | Pre-Post comparison (28 days)
  Number of participants with clinically meaningful change in PAC-QoL (reduction of >0.5 or >1.0 point).
  A validated questionnaire consisting of 28 items to measure the impact of constipation on a patient's quality of life.
Participant Compliance | Pre-Post comparison (28 days)
  Number of participants completing >75% of breath gas measurements and bowel diary submissions with OMED device.
  The OMED Health Breath Analyzer is used for breath gas readings at 4 intervals during the day. The bowel diary recorded daily on paper throughout the study capturing movements, symptoms and any medication
Whole Gut Transit Time (ATMO) | Pre-Post comparison (28 days)
  Change in whole gut transit time measured by ATMO capsule
  ATMO capsule is an ingestible electronic medical device measuring gastrointestinal (GI) transit time and environmental conditions as it moves through the digestive tract.
Whole Gut Transit Time (Blue-dye) | Pre-Post comparison (28 days)
  Change in whole gut transit time measured by Blue dye transit study baseline period to treatment period.
  Participants are required to consume a Zoe blue cookie the following morning after both visits 2 and 3. Participants then report when the blue food colour is visible in their stool, checking every time they pass a bowel movement.
Small Bowel Transit Time (ATMO) | Pre-Post comparison (28 days)
  Change in small bowel transit time measured by ATMO capsule
  ATMO capsule is an ingestible electronic medical device measuring gastrointestinal (GI) transit time and environmental conditions as it moves through the digestive tract.
Large Bowel Transit Time (ATMO) | Pre-Post comparison (28 days)
  Change in large bowel transit time measured by ATMO capsule
  ATMO capsule is an ingestible electronic medical device measuring gastrointestinal (GI) transit time and environmental conditions as it moves through the digestive tract.
Gastrointestinal Symptom Rating Scale (GSRS) | Pre-Post comparison (28 days)
  Mean change in GSRS score
  A validated questionnaire consisting of 15items to assess range of GI symptoms. Scored using a seven-graded Likert scale, where 1 represents the most positive option and 7 the most negative one.
Stool form comparison | Pre-Post comparison (days 1-14 compared to days 29-42)
  Average stool type recorded in two week baseline compared to average stool type recorded final two weeks of treatment period. Measured using the bristol stool chart reported in bowel habit diary.
Stool frequency comparison | Pre-Post comparison (days 1-14 compared to days 29-42)
  Average stool frequency recorded in two week baseline compared to average stool type recorded final two weeks of treatment period reported in bowel habit diary.
Hydrogen and methane production | Pre-Post comparison (days 1-14 compared to days 15-42)
  Assessment of longitudinal hydrogen and methane production during baseline and treatment periods. Recorded by OMED device 4x daily
Global PAC-SYM | Pre-Post comparison (28 days)
  Comparison of global PAC-SYM score from baseline period to treatment period.
Inidividual PAC-SYM | Pre-Post comparison (28 days)
  Comparison of individual PAC-SYM symptom scores from baseline period to treatment period.
Straining | Pre-Post comparison (days 1-14 compared to days 15-42)
  Self reported straining recorded in two week baseline compared to self reported straining during treatment period reported in bowel habit diary.
Sense of complete evacuation | Pre-Post comparison (days 1-14 compared to days 15-42)
  Self reported sense of complete evacuation recorded in two week baseline compared to self reported Sense of complete evacuation during treatment period reported in bowel habit diary.
Time taken for evacuation | Pre-Post comparison (days 1-14 compared to days 15-42)
  Self reported time taken for evacuation recorded in two week baseline compared to self reported time taken for evacuation during treatment period reported in bowel habit diary.
Rescue Medication | Pre-Post comparison (days 1-14 compared to days 15-42)
  Self reported use of rescue medication recorded in two week baseline compared to self reported use of rescue medication during treatment period reported in bowel habit diary.

CONTACTS AND LOCATIONS:
Locations (1):
- The Functional Gut Clinic, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided